CLINICAL TRIAL: NCT00002213
Title: A Phase II Study Evaluating the Safety and Antiviral Activity of Combination Therapy With 1592U89, 141W94 and DMP 266 in HIV-1 Infected Subjects With Detectable HIV-1 Plasma RNA Despite Treatment With a Protease Inhibitor Containing Regimen
Brief Title: The Safety and Effectiveness of 1592U89 Plus 141W94 Plus DMP 266 in Patients With HIV Who Developed a Resistance to Protease Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 264F; CNAA2007
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-03

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Antiviral Agents; HIV Protease Inhibitors; RNA, Viral; VX 478; Anti-HIV Agents; abacavir; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — abacavir; amprenavir; efavirenz

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Efavirenz

SUMMARY:
The purpose of this study is to see if it is safe and effective to give 1592U89 plus 141W94 plus DMP 266 to patients with HIV who have developed resistance to indinavir, ritonavir, saquinavir, or nelfinavir after at least 20 weeks of protease inhibitor treatment. This study also examines how long this combination therapy is effective before patients develop resistance to it.

DETAILED DESCRIPTION:
This is a multicenter, open-label study. A total of 80 patients are treated on this study and include:

At least 30 patients with a viral burden of 500 - 40,000 copies/ml. At least 30 patients with a viral burden greater than 40,000 copies/ml. At least 20 patients with less than 1 year total prior treatment with nucleoside reverse transcriptase inhibitors (NRTIs).

All patients receive self-administered, combination antiretroviral therapy for 48 weeks, as follows:

1592U89 plus 141W94 plus DMP 266.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Hematologic supportive therapy with GM-CSF, G-CSF, or erythropoietin.
* Drugs that may interact with CYP3A4, that should be used with caution including (but not limited to):
* alprazolam, carbamazepine, codeine, cimetadine, clarithromycin, dapsone, diazepam, diltiazem, erythromycin, estrogens, fluvastatin, glucocorticoids, imipramine, itraconazole, ketoconazole, lidocaine, lovastatin, nifedipine, phenobarbital, phenytoin, quinidine, rifabutin, simvastatin, and warfarin.
* Detoxification treatment including opiate agonists (methadone, buprenorphine, etc.):
* Patients currently receiving this treatment should be enrolled only if stable on this therapy.

Patients must have:

* HIV-1 infection (all CDC clinical categories allowed).
* HIV-1 RNA greater than 500 copies/ml when measured on 1 occasion within 14 days of study drug administration.
* Signed, informed consent from parent or legal guardian for those patients under 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malabsorption syndrome or other gastrointestinal dysfunction that may interfere with drug absorption or render the patient unable to take oral medication.
* Active AIDS-defining opportunistic infection or disease that is likely to preclude the patient from study participation.
* Serious medical conditions such as diabetes, congestive heart failure, cardiomyopathy, or other cardiac dysfunction that, in the opinion of the investigator, would compromise the safety of the patient.

Concurrent Medication:

Excluded:

* Immunomodulating agents, e.g., corticosteroids, interleukins, thalidomide, anti-cytokine agents and interferons.
* Cytotoxic chemotherapeutic agents (except local treatment for Kaposi's sarcoma).
* Anti-oxidants.
* Foscarnet therapy or therapy with other agents with documented activity against HIV-1 in vitro.
* Medications that interact with 141W94:
* terfenadine, astemizole, cisapride, triazolam, midazolam, and ergotamine/dihydroergotamine-containing regimens.
* Vitamin E supplements.
* Other investigational treatments (treatments available through Treatment IND or other expanded access mechanism evaluated on an individual basis).

Concurrent Treatment:

Excluded:

Anticipated need for radiation therapy (with the exception of local treatment for Kaposi's sarcoma).

Patients with the following symptoms and conditions are excluded:

* History of clinically relevant hepatitis within the previous six months.
* History of lymphoma.

Prior Medication:

Excluded:

* Cytotoxic chemotherapeutic agents within 30 days of study drug administration or an anticipated need for such treatment within the next 48 weeks (with exception of local treatment for Kaposi's sarcoma).
* Investigational HIV-1 vaccine trial and receipt of a dose of vaccine within the past 3 months.
* Immunomodulating agents such as systemic corticosteroids, interleukins, or interferons within 30 days of study drug administration.
* Exposure to the investigational agents 1592U89, 141W94, or DMP 266 (Sustiva).

Prior Treatment:

Excluded:

Radiation therapy.

Required:

* Treatment with at least 1 of the following protease inhibitors (PIs) for a minimum of 20 weeks prior to screening:

indinavir, ritonavir, saquinavir, and/or nelfinavir.

* Treatment with the same combination of PIs for the most recent 12 weeks and up through entry on study (Day 1).

Active alcohol or illicit drug use that is likely to interfere with dosing schedule compliance and protocol evaluations.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - East Bay AIDS Ctr, Berkeley, California
  - Kraus Med Partners, Los Angeles, California
  - Northwestern Univ Med School AIDS Treatment Unit, Chicago, Illinois
  - Niaid / Nih, Bethesda, Maryland
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Saint Vincents Hosp / AIDS Ctr / 4th Floor, New York, New York
  - Univ of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Univ Int Med Assoc Inc / Holmes Hosp / U of Cincinnati, Cincinnati, Ohio
  - The Miriam Hosp, Providence, Rhode Island